CLINICAL TRIAL: NCT05398458
Title: Management of a Giant Lymphocele Following Varicose Vein Surgery - A Case Report
Status: Completed | Type: Observational
Sponsor: Bahria International Hospital (Unknown)
Responsible Party: Principal Investigator, Dr Noshi Bibi, Noshi Bibi, Bahria International Hospital
Other Study IDs: BIH
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Lymphocele; Varicose Veins
Keywords: Lymphocele, Varicose Vein, Gracilis Muscle, Sclerotherapy.
MeSH Terms: conditions — Lymphocele; Varicose Veins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Lymphocele excision and space obliterated by pedicle Gracilis muscle only flap — By this procedure it has helped in reduction and complete resolution of the lymphocele with no recurrence in the past 2 years

SUMMARY:
A 48-year-old female presented to the plastic surgery outpatient department (OPD) with a history of painful, progressive swelling of the right groin and medial aspect of the right thigh for 4 months. After investigation, it was diagnosed as a giant lymphocele. A pedicled gracilis muscle flap was used to reconstruct and obliterate the cavity. There was no recurrence of the swelling. : Lymphocele is a common complication after extensive vascular surgeries. In the unfortunately case of its development, prompt intervention must be done to prevent its growth and ensuing complications.

ELIGIBILITY:
Inclusion Criteria: diagnosed case of lymphocele -

Exclusion Criteria: none

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: post varicose vein surgery ,patient developed lymphocele in right thigh
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Management of a Giant Lymphocele Following Varicose Vein Surgery - A Case Report | 2 year
  Complete resolution of lymphocele

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria iInternational Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided